CLINICAL TRIAL: NCT05303714
Title: Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) in Multimodal Therapy for Patients with Oligometastatic Peritoneal Gastric Cancer: a Randomized Multicenter Phase III Trial: PIPAC_VEROne
Brief Title: PIPAC in Multimodal Therapy for Patients with Oligometastatic Peritoneal Gastric Cancer
Acronym: PIPAC_VEROne
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Francesco Casella, Francesco Casella MD, Principal Investigator, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIPAC_VEROne
Record Dates: First submitted 2022-02-15; First posted 2022-03-31 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-08

CONDITIONS: Oligometastatic Gastric Adenocarcinoma
MeSH Terms: interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (FOLFOX) (Active Comparator): Patients randomized in the Arm A will undergo to 6 courses of systemic chemotherapy according to FOLFOX regimen, after these six courses of chemotherapy, radiologic restaging (CT scan) as well as a second staging laparoscopy will be performed. If a Progression Disease will be detected, the patient will end the trial and will undergo to II line chemotherapy regimen. If a stable disease or a partial response will be documented, after a multidisciplinary discussion, patient will undergo to either further 6 courses of chemotherapy or to cytoreductive surgery plus HIPEC.
  Interventions: Combination Product: FOLFOX and PIPAC
- Arm B (FOLFOX and PIPAC) (Experimental): Patients randomized in the ARM B will undergo to 6 courses of systemic chemotherapy (FOLFOX regimen) plus PIPAC every two cycles of chemo (Fig.1). At least seven days should last between each PIPAC and the next chemotherapy course, and at least 14 days should last between the chemotherapy course and the next PIPAC. After six courses of chemotherapy and 3 PIPACs procedure, a radiologic restaging (CT scan) as well as a laparoscopic reassessment will be performed. If a Progression Disease will be detected, the patient will end the trial and will undergo to II line chemotherapy regimen. If a stable disease or a partial response will be documented, patient will be treated with cytoreductive surgery plus HIPEC.
  Interventions: Combination Product: FOLFOX and PIPAC

INTERVENTIONS:
Combination Product: FOLFOX and PIPAC — A minilaparotomy is performed in the midline. A 5 mm balloon trocar is inserted under "finger protection" in the right side and the fascia of the minilaparotomy is closed. The abdomen is insufflated with CO2 and a second 10-12mm trocar is introduced under videoscope control in upper left side. Ascites volume is documented and removed sending a sample for cytological examination, an accurate exploratory laparoscopy is performed, possibly placing an additional 5 or 10-12 mmHg trocar, the Peritoneal Cancer Index is calculated. Multiple biopsies are performed in different abdominal quadrants. A nebulizer CAPNOPEN© is inserted into the upper left side trocar and fixed with a 45° angle. The drugs (Cisplatin 10.5 mg/m2 body surface in 150 mL; Doxorubicin 2.1 mg/m2 body surface in 50 mL) are then injected through remote control with a flow rate of 0.7 mL/sec with a pressure of 200 psi. After an aerosol exposure phase of 30min, the aerosol is evacuated via a closed waste system.

SUMMARY:
Peritoneal Carcinomatosis is the most frequent site of metastases observed in patients with gastric cancer. Current standard treatment for these patients is palliative systemic chemotherapy, but the prognosis is very poor. Cytoreductive surgery (CRS) combined with hyperthermic intraperitoneal chemotherapy (HIPEC) resulted in long-term benefits in selected patients with limited peritoneal involvement. Indeed, among patients with Peritoneal Carcinomatosis, a distinctive subset is oligometastatic disease which is characterized by low metastatic burden. PIPAC is a recent technique of intraperitoneal chemotherapy that can be used in combination with systemic chemotherapy with promising results for patients with PM from gastric cancer. The role of PIPAC in multimodal treatment path for oligometastatic gastric cancer should be investigated in clinical trials. PIPAC VER-One is a prospective, randomized, multicenter phase III clinical trial with two arms that aims to evaluate the effectiveness of the use of PIPAC in combination with systemic chemotherapy in patients with Gastric Cancer and synchronous positive peritoneal cytology and/or limited peritoneal metastases (PCI ≤ 6). Patients will be randomized into two arms: arm A (control) treated with the current standard that is systemic chemotherapy only and Arm B (experimental) treated with a bidirectional scheme including PIPAC and systemic chemotherapy (1 PIPAC every 2 systemic chemotherapy cycles). Primary endpoint is the Secondary Resectability Rate. Secondary endpoints are: Overall Survival, Progression Free Survival, Disease Free Survival, histological response assessed both on primary tumor and peritoneal lesions, Quality of Life, complication rate (CTCAE v5), incremental cost-effectiveness ratios (ICER).

DETAILED DESCRIPTION:
This is a prospective, open label, randomized multicenter phase III clinical study that aims to evaluate the effects of PIPAC combined with systemic chemotherapy vs. intravenous systemic chemotherapy alone on patients with gastric cancer and synchronous positive peritoneal cytology and/or limited peritoneal metastasis (PCI ≤ 6). Patients will be randomly assigned in a 1:1 ratio to Arm A: intravenous chemotherapy (FOLFOX) vs. Arm B: intravenous chemotherapy (FOLFOX) plus PIPAC with cisplatin and doxorubicin.

Patients eligible for the trial must have performed: diagnostic upper intestinal endoscopy with biopsies, thoraco-abdominal-pelvic CT scan, laboratory exams: serum CEA, CA19.9, hemoglobin, leukocytes, neutrophils, platelets, glycemia, AST, ALT, LDH, total bilirubin, alkaline phosphatase, serum albumin, total protein, plasmatic APTT, PT, creatinine clearance and serum creatinine and pregnancy serological test.

Patients should undergo to staging laparoscopy in one of the participating centers to define the peritoneal involvement. After that peritoneal metastasis will be confirmed by cytological/histopathological final examination and after receiving the written informed consent, patient will be randomized.

Once the inclusion and exclusion criteria are confirmed, each patient will be randomized in a 1:1 ratio (Chemotherapy alone vs chemotherapy plus PIPAC) to blocks of 14 using a centralized randomization list, stratified by center. Randomization list will be managed by the Medical Epidemiology and Statistics Unit, Department of Diagnostics and Public Health of the University of Verona. This list will be built using the Biostatistics Unit of the University of Verona using software (www.randomizer.org) Patients randomized in the Arm A will undergo to 6 courses of systemic chemotherapy according to FOLFOX regimen, after these six courses of chemotherapy, radiologic restaging (CT scan) as well as a second staging laparoscopy will be performed. If a Progression Disease will be detected, the patient will end the trial and will undergo to II line chemotherapy regimen. If a stable disease or a partial response will be documented, after a multidisciplinary discussion, patient will undergo to either further 6 courses of chemotherapy or to cytoreductive surgery plus HIPEC.

Patients randomized in the ARM B will undergo to 6 courses of systemic chemotherapy (FOLFOX regimen) plus PIPAC every two cycles of chemo. At least seven days should last between each PIPAC and the next chemotherapy course, and at least 14 days should last between the chemotherapy course and the next PIPAC. After six courses of chemotherapy and 3 PIPACs procedure, a radiologic restaging (CT scan) as well as a laparoscopic reassessment will be performed. If a Progression Disease will be detected, the patient will end the trial and will undergo to II line chemotherapy regimen. If a stable disease or a partial response will be documented, patient will be treated with cytoreductive surgery plus HIPEC.

A minilaparotomy of 3 cm is performed, usually in the midline. Then, a 5 or a 10-12 mm balloon trocar is inserted under "finger protection" usually in the right side and the fascia of the minilaparotomy, is then closed. The abdomen is insufflated with CO2 and tightness is controlled with saline solution in the minilaparotomy. CO2-bubbling documents incomplete closure. A second 10-12mm trocar is then introduced safely under videoscope control usually in upper left side. Ascites volume is documented, and ascites is removed sending a sample for cytological examination, an accurate exploratory laparoscopy is performed, possibly placing an additional 5 or 10-12 mmHg trocar in an area not affected by adhesions or disease, the Peritoneal Cancer Index is calculated. Multiple biopsies are performed in different abdominal quadrants during the first procedure and all following procedures to ascertain tumor regression grade. Then, a nebulizer CAPNOPEN© is connected to an intravenous high-pressure injector and inserted into the upper left side trocar and fixed with a 45° angle to the underlying peritoneum to allow a better spatial drug distribution pattern and a greater spraying distance between the nozzle head and the underlying small bowel peritoneum compared to the that obtained with a perpendicular nozzle position.

The liquid chemotherapeutic drugs (Cisplatin 10.5 mg/m2 body surface in a total of 150 mL NaCl 0.9 %; Doxorubicin 2.1 mg/m2 body surface in a total of 50 mL NaCl 0.9 %) are then injected through remote control with a flow rate of 0.7 mL/sec with a maximum operating pressure of 200 psi (13 bar) into the constant capnoperitoneum of 12 mm Hg. After an aerosol exposure phase of 30min, the aerosol is evacuated via a closed aerosol waste system. Finally, trocars are retracted, and laparoscopy ended. No drainage of the abdomen is applied.

FOLFOX regimen systemic chemotherapy will be administered to each patient in both arms.

Arm A will receive only systemic chemotherapy according to this scheme: Oxaliplatin 85 mg/m2, d1, over 2 h, Leucovorin 400 mg/m2, d1 i.v. over 2 h, 5-FU 400 mg/m2 in bolus and 5-FU 2.400mg/m2, d1, i.v. over 46 h. Arm B will be treated with systemic chemotherapy plus PIPAC procedure according to this scheme (Fig.1): PIPAC with Cisplatin 10,5 mg/m2 and Doxorubicin 2,1 mg/m2; chemotherapy with the same way of Arm A. At least seven days should last between each PIPAC and the next chemotherapy cycle, and at least 14 days should last between the chemotherapy cycle and the following PIPAC procedure.

Secondary Resectability Rate (%) evaluated as the rate of patients of the two arms that get radical intent surgery (cytoreductive surgery and HIPEC).

According to the current literature, considering a resectability rate of 50%9 for patients undergoing chemotherapy alone (arm A) and 80% in the experimental arm (arm B), the investigators need 88 patients (44 per group) to achieve 80% potency by performing an exact bidirectional Fisher test with an alpha of 5%.

Expecting a dropout rate of 10% it will be necessary to recruit 98 patients, 49 for each arm. A very similar recruitment capacity is envisaged in the different centers.

The enrollment of patients will last about three and a half years from the date of approval. An enrollment of about 30 patients per year is expected in the 7 centers involved. If the enrollment is lower than expected, up to 10 centers will be recruited and the enrollment period will be extended. These latter changes will be the subject of any future substantial amendment to the current study protocol.

Patients will be involved in the study from the time of enrollment, the duration of treatment (from a minimum of 3 months to a maximum of 6 months) and for the next 3 years of follow-up.

The clinical trial will last a total of six and a half years. The end of data collection coincides with the achievement of a three-year follow-up for the last patient enrolled. An additional year will be needed for the analysis of the data and the publication of the results.

ELIGIBILITY:
Inclusion Criteria:

* Primary resectable gastric cancer with positive peritoneal cytology and/or low burden peritoneal metastases (PCI ≤6) confirmed by laparoscopy
* Signature of written informed consent
* ECOG PS 0-1

Exclusion Criteria:

* Extraperitoneal metastases
* PCI >6
* Gastro-esophageal junction tumor of esophageal relevance (Siewert I-II)
* Previous allergic reactions to cisplatin or doxorubicin
* Hemorrhagic or occlusive manifestation of the primary tumor with palliative surgery needed
* ASA IV
* Positivity for EBV, MSI and HER2 on diagnostic biopsies
* Pregnancy and breastfeeding
* Contraindication to any drug contained in the chemotherapy regimen
* Hepatic impairment (AST/ALT> 3 times normal values, ALT>3 times normal values, Bilirubin>1.5 normal values)
* Ischemic/hemorrhagic stroke in the last 6 months
* Acute myocardial infarction in the last 6 months
* Moderate/severe heart failure (NYHA III-IV)
* Leukopenia< 2,000/μl
* Thrombocytopenia < 100,000/μl
* Active hepatitis B or C
* HIV infection
* Creatinine clearance less than 30 ml/min

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Secondary Resectability Rate (percent) | Three and a half years
  The rate of patients of the two arms that get radical intent surgery (cytoreductive surgery and HIPEC)

SECONDARY OUTCOMES:
OS | Three and a half years
  Overall Survival
PFS | Three and a half years
  Progression-Free Survival
DRS | Three and a half years
  Disease-related survival
PRGS | Three and a half years
  Peritoneal Regression Grade Score: Grade 1 complete response; Grade 2 major response; Grade 3 minor response; Grade 4 no response.
TRG | Three and a half years
  Tumor Regression Grading according Mandard: TRG 1 complete regression; TRG 2 presence of rare residual cancer cells scattered through the fibrosis; TRG 3 was increase in the number of residual cancer cells, but fibrosis still predominated; TRG 4 residual cancer outgrowing fibrosis; and TRG 5 absence of regressive changes.
  Tumor Regression Grading according Becker: Grade 1, complete (Grade 1a) or subtotal tumor regression (< 10% residual tumor per tumor bed; Grade 1b); Grade 2, partial tumor regression (10-50% residual tumor per tumor bed), and Grade 3, minimal or no tumor regression (> 50% residual tumor per tumor bed).
Quality of Life according EORTC QLQ-C30 | Three and a half years
  The EORTC Core Quality of Life questionnaire (EORTC QLQ-C30) is designed to measure cancer patients' physical, psychological and social functions. The questionnaire is composed of multi-item scales and single items.
Complication rate | Three and a half years
  CTCAE and Clavien-Dindo

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Casella, Principal Investigator — General and Upper GI Surgery, University of Verona
Locations (1):
- AOUI Verona, Verona, Italy

REFERENCES:
- See also: University of Verona — http://www.univr.it